CLINICAL TRIAL: NCT05331898
Title: The Effect Of Rational Drug Use Education Given To Parents On Parental Attitudes
Brief Title: Rational Drug Use Education Parental Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/502
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Disorder
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): increase the rational drug use of the parents.
  Interventions: Behavioral: Education
- control (No Intervention): PARENTS CANNOT USE RATIONAL MEDICATION ON THEIR CHILDREN

INTERVENTIONS:
Behavioral: Education — the education given increased the rational drug use of the parents.
  Arms: Education Group

SUMMARY:
The study aims to examine the effect of rational drug use education given to parents on parental attitudes. The pretest-posttest randomized controlled experimental study was carried out in Erzurum between June 2020 and September 2021. The study's population comprised parents with children aged 0 to 12 who were registered at an Erzurum FHC. The study sample consisted of 100 parents who came to the FHC on the specified dates and matched research criteria. "Parent Introductory Information Form", "Parental Attitude Scale for Rational Drug Use (PASRDU)" and "Rational Drug Use Education" were used to collect research data.

DETAILED DESCRIPTION:
Type of the Research The study was conducted as a randomized controlled trial with a pretest-posttest design.

Place and Time of the Research The research was conducted between June 2020 and September 2021 in a Family Health Center (FHC) in Erzurum.

Population and Sample of the Research The study's population comprised parents with children aged 0 to 12 who were registered at an Erzurum FHC. Using the probabilistic sampling method, the study sample consisted of 100 parents who came to the FHC on the specified dates and matched the research criteria. Power analysis was used to determine the sample size in the study using the G.Power 3.1.9.2 application. In the power analysis, it was determined that 104 parents should be reached, 52 parents in the experimental group and 52 parents in the control group, with a 95% confidence interval, 80% theoretical power, and 0.5 impact power. At this point, 2 experimental and 2 control parents who did not want to participate in the study were removed from the study, bringing the total number of participants to 100 (50 experimental, 50 control).

Inclusion criteria for the study;

* Being a 0-12 age group child
* Being literate
* Not having any communication problems
* Previous drug use for the child. Data Collection Tools "Parent Introductory Information Form", "Parental Attitude Scale for Rational Drug Use" and "Rational Drug Use Education" were used to collect research data.

Parent Introductory Information Form: In this form, which was prepared by the researcher based on the literature, there are 13 questions in total about age, gender, place of residence of the parents, family type, social security, socioeconomic level, educational status, and occupation, the number of children aged 0-12, the presence of children with chronic diseases, where they most often apply for drug treatment when their child is sick, and the most frequently non-prescribed drugs.

Parental Attitude Scale for Rational Drug Use (PASRDU): It was developed in 2018. The scale consists of 2 sub-dimensions and 40 items. The sub-dimensions of the scale "Correct and Conscious Use" consist of 29 items and "Effective and Safe Use" consists of 11 items. PASRDU is a 5-point Likert-type scale consisting of five questions with the answers "(1) strongly disagree, (2) disagree, (3) indecisive, (4) agree, (5) strongly agree". While 12 of the 40 items in the scale were negative (16,30,31,32,33,34,35,36,37,38,39,40) statements, 28 items consisted of positive statements. The negative items were reverse-scored. The higher the score obtained from the scale, the higher the positive attitude of parents towards rational drug use.

Rational Drug Use Education: An education booklet was created by the researchers based on the literature. What is a drug? What is rational drug use? What are the benefits of rational drug use? What are the principles of rational drug use? What is irrational drug use? What are the main effects of irrational drug use? What are the problems of irrational drug use? Who makes up the rational drug use team? What are the most common errors mothers make when giving their children drugs? What should be known about rational drug use? What should we pay attention to when giving a drug to children? These are some of the questions it contains.

Data Collection Control Group: Initially, control group data were collected. In the first interview, pre-test data were collected by applying the "Parent Introductory Information Form" and "Parental Attitude Scale for Rational Drug Use". It took roughly 15-20 minutes to complete the forms. No education was provided. Covid-19 precautions were taken while collecting data. One month after the pre-test application, the post-test was applied. Post-test data were collected by the telemonitoring method.

Experimental Group: In the first interview, pre-test data were collected by applying the "Parent Introductory Information Form" and "Parental Attitude Scale for Rational Drug Use. It took roughly 15-20 minutes to complete the forms. A PowerPoint presentation developed by the researcher was used to provide rational drug use training. The parents were given the prepared education booklet so that they may utilize it whenever they required it. Covid-19 precautions were taken while collecting data. One month after training, posttest data were collected. Telemonitoring method was used to collect post-test data.

Variables of the Research Dependent Variable: "Parental Attitude Scale for Rational Drug Use" score averages of parents Independent Variable: "Rational Drug Use" education given to parents Control Variable: Introductory characteristics of parents Evaluation of the Data Statistical analysis of the research data was evaluated using the SPSS 22.0 (Statistical Package for Social Science) package program. Continuous variables were given as mean±standard deviation and categorical variables as numbers and percentages. The student's t-test was used for two-group comparisons of normally distributed quantitative data. A Paired-Sample t-test was used to compare the normally distributed scale scores before and after education. Additionally, differences between categorical variables were analyzed by Chi-square analysis. The significance level was set as p˂0.05.

Ethical Principles of the Research Ethical approval of the Ethics Committee was obtained for the study. The research group's parents were informed about the study's purpose, their questions were answered, and their verbal and written consents were obtained. The parents were informed that the information they supplied would be kept private and would not be shared with anyone else and that they had the right to withdraw from the study at any time. Since the use of the human phenomenon requires the protection of individual rights, the relevant ethical principles "Principle of Informed Consent", "Principle of Volunteering" and "Principle of Protection of Confidentiality" were fulfilled in the research.

ELIGIBILITY:
Inclusion Criteria:

* Being a 0-12 age group child
* Being literate
* Not having any communication problems
* Previous drug use for the child.

Exclusion Criteria:

* 0-12 age group without children
* Being illiterate
* Having communication problems
* The child does not use drugs.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Parental Attitude Scale for Rational Drug Use | 15 MONTHS
  It was developed in 2018. The scale consists of 2 sub-dimensions and 40 items. The sub-dimensions of the scale "Correct and Conscious Use" consist of 29 items and "Effective and Safe Use" consists of 11 items. PASRDU is a 5-point Likert-type scale consisting of five questions with the answers "(1) strongly disagree, (2) disagree, (3) indecisive, (4) agree, (5) strongly agree". While 12 of the 40 items in the scale were negative (16,30,31,32,33,34,35,36,37,38,39,40) statements, 28 items consisted of positive statements. The negative items were reverse-scored. The higher the score obtained from the scale, the higher the positive attitude of parents towards rational drug use.

CONTACTS AND LOCATIONS:
Overall Officials: ARZU SARIALİOĞLU, PHD, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTICLE IS INTENDED TO BE SHARED AFTER IT IS PUBLISHED